CLINICAL TRIAL: NCT01982942
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Activity of Ibudilast (MN-166) in Subjects With Progressive Multiple Sclerosis
Brief Title: Safety, Tolerability and Activity Study of Ibudilast in Subjects With Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN102 SPRINT - MS; 1U01NS082329-01A1 (NIH); RG 4778-A-6 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibudilast (Experimental): Subjects will receive up to 100 mg/d ibudilast for 96 weeks.
  Interventions: Drug: ibudilast
- Placebo Oral Capsule (Placebo Comparator): Subjects will receive placebo for 96 weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ibudilast — Subjects randomly assigned to the ibudilast (MN-166) cohort will receive up to 100 mg/day for 96 weeks.
  Other Names: MN-166
  Arms: ibudilast
Drug: Placebo oral capsule — Subjects randomly assigned to the placebo cohort will receive placebo oral capsule for 96 weeks.
  Arms: Placebo Oral Capsule

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the safety, tolerability and activity of ibudilast administered twice daily over a 96 week period in subjects with primary or secondary progressive multiple sclerosis who are currently untreated with long-term MS disease modifying therapy (DMT) or who are receiving either glatiramer acetate (GA) or interferon beta-1, any formulation (IFNβ-1A [Avonex, Rebif] or IFNβ-1B [Betaseron, Extavia]). Study drug or placebo will be administered to a total of 250 male and female subjects from 21 to 65 years old, inclusive, in two treatment groups. Randomization of subjects will be stratified by disease status (primary progressive multiple sclerosis or secondary progressive multiple sclerosis) and immunomodulating therapy status: current use of immunomodulating therapy or no current use of immunomodulating therapy.

The study will consist of a screening phase (up to 30 days) followed by a treatment phase (96 weeks) and a follow-up visit (1 month post Week 96 visit). Following the screening phase, subjects who continue to meet entry criteria will be randomly assigned to 1 of 2 treatment groups: doses up to ibudilast 100 mg/day or matching-placebo in a 1:1 ratio. Study drug will be administered twice daily (BID), e.g., ibudilast 50 mg or placebo taken in the morning and evening).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained and willing and able to comply with the protocol in the opinion of the Investigator.
* Male or female subjects ages 21 to 65, inclusive
* Confirmed diagnosis of SPMS or primary progressive multiple sclerosis (PPMS) according to 2010 International Panel Criteria
* Typical MS lesions on MRI according to Swanton's MRI Criteria (at least one lesion in two or more of the following regions: periventricular, juxtacortical, infratentorial [brainstem/cerebellum], spinal cord)
* EDSS 3.0-6.5, inclusive
* Clinical evidence of disability progression in the preceding two years, as measured by any of the following (excluding progression during clinical relapses):

  * worsening overall EDSS of at least 0.5 points (may be assessed retrospectively but cannot be during a clinical relapse) or
  * 20% worsening in 25-foot walk (25-FW) or
  * 20% worsening in 9-hole peg test (9-HPT) in either hand
* Existing multiple sclerosis pharmacotherapy status may include interferon-beta or glatiramer acetate or none (i.e. untreated).
* Females of child-bearing potential must have a negative serum ß-hCG at screening and must be willing to use appropriate contraception (as defined by the investigator) for the duration of study treatment and 30 days after the last dose of study treatment.
* Males should practice contraception as follows: condom use and contraception by female partner.
* Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening, as defined by the investigator.
* Subject is willing and able to comply with the protocol assessments and visits, in the opinion of the study nurse/coordinator and the Investigator.

Exclusion Criteria:

* Progressive neurological disorder other than SPMS or PPMS
* Relapse and/or systemic corticosteroid steroid treatment for multiple sclerosis within 3 months of screening. Inhaled or topical steroids are allowed.
* Current use of intermittent systemic corticosteroids (i.e., monthly or bimonthly intravenous methylprednisolone)
* Use of oral immunosuppressants (e.g. azathioprine, methotrexate, cyclosporine, teriflunomide [Aubagio®]) within 6 months of screening
* Use of mitoxantrone, natalizumab, or IVIg within 6 months of screening
* Use of fingolimod or dimethyl fumarate [Tecfidera®] within 3 months of screening
* Use of rituximab or other B-cell therapy within 12 months of screening
* Current use of other MS disease-modifying therapies (DMTs) besides glatiramer acetate, IFNβ-1 (any formulation), and the above listed medications.
* Current use of cimetidine, cyclosporine, dronedarone, lopinavir, probenecid, quinidine (including Neudexta), ranolazine, rifampin, ritonavir, or tipranavir.
* Clinically significant cardiovascular disease, including myocardial infarct within last 6 months, unstable ischemic heart disease, congestive heart failure or angina
* Resting pulse < 50 bpm, sinoatrial (SA) or atrioventricular (AV) block, uncontrolled hypertension, or QTcF > 450 ms
* Clinically significant pulmonary conditions, including severe chronic obstructive pulmonary disease (COPD), fibrosis, or tuberculosis
* Evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation including ALP > 1.5x ULN; ALT or AST > 2x ULN; GGT > 3x ULN
* Immune system disease (other than multiple sclerosis and autoimmune thyroid disease)
* History of stomach or intestinal surgery or any other condition that could interfere with or is judged by the Investigator to interfere with absorption, distribution, metabolism, or excretion of study drug.
* Any significant laboratory abnormality which, in the opinion of the Investigator, may put the subject at risk and with the following laboratory abnormalities at screening:

  * Creatinine: females > 0.95 mg/dL; males > 1.17 mg/dL
  * WBCs < 3,000 mm3
  * Lymphocytes < 800 mm3
  * Platelets < 90,000 mm3
* History of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* History of HIV (human immunodeficiency virus), clinically significant chronic hepatitis, or other active infection.
* Subject currently has a clinically significant medical condition (other than MS) including the following: neurological, psychiatric, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular (including uncontrolled hypertension), gastrointestinal, urological disorder, or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if, in the judgment of the Investigator, they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Safety Monitor should be consulted.

* Subjects with moderate to severe depression as determined by the Beck Depression Inventory-Fast Screen (BDI-FS).
* Subject has a history of alcohol or substance abuse (DSM-IV-TR criteria) within 3 months prior to screening or alcohol or substance dependence (DSM-IV-TR criteria) within 12 months prior to screening. The only exceptions include caffeine or nicotine abuse/dependence.
* Subject has poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator.
* Subject is currently participating, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent.
* Subject is unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator, or was planning to relocate during the study.
* Subject is unable to undergo MRI imaging because of having an artificial heart valve, metal plate, pin, or other metallic objects (including gun shots or shrapnel) in their body or is unable to complete all the five MRI scans required for this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Fox, MD, FAAN, Principal Investigator — The Cleveland Clinic
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis, Davis, California
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine in St Louis, St Louis, Missouri
  - University at Buffalo, The State University of New York, Buffalo, New York
  - Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University at Stony Brook, The State University of New York, Stony Brook, New York
  - University at Upstate, The State University of New York, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Department of Neurology, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Charlottesville, Charlottesville, Virginia
  - Swedish Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Derived] Krijnen EA, Bruijn AM, Eloyan A, Schoonheim MM, Fox RJ, Klawiter EC. Evaluation of cortical pathology in primary-progressive multiple sclerosis: a post hoc analysis of the SPRINT-MS trial. BMJ Neurol Open. 2026 Jan 5;8(1):e001335. doi: 10.1136/bmjno-2025-001335. eCollection 2026. PMID 41509523
- [Derived] Novak A, Harvey T, Wojdala A, Teunissen C, Fox R. Effect of Ibudilast vs Placebo on GFAP and Contactin levels in a phase 2 clinical trial in progressive multiple sclerosis. Neurol Open Access. 2025 Dec;1(4):10.1212/wn9.0000000000000040. doi: 10.1212/wn9.0000000000000040. Epub 2025 Nov 21. PMID 41342004
- [Derived] Singh V, Zheng Y, Ontaneda D, Mahajan KR, Holloman J, Fox RJ, Nakamura K, Trapp BD. Disability independent of cerebral white matter demyelination in progressive multiple sclerosis. Acta Neuropathol. 2024 Aug 31;148(1):34. doi: 10.1007/s00401-024-02796-w. PMID 39217272
- [Derived] Nakamura K, Zheng Y, Mahajan KR, Cohen JA, Fox RJ, Ontaneda D. Effect of ibudilast on thalamic magnetization transfer ratio and volume in progressive multiple sclerosis. Mult Scler. 2023 Sep;29(10):1257-1265. doi: 10.1177/13524585231187289. Epub 2023 Aug 3. PMID 37537928
- [Derived] Bermel RA, Fedler JK, Kaiser P, Novalis C, Schneebaum J, Klingner EA, Williams D, Yankey JW, Ecklund DJ, Chase M, Naismith RT, Klawiter EC, Goodman AD, Coffey CS, Fox RJ. Optical coherence tomography outcomes from SPRINT-MS, a multicenter, randomized, double-blind trial of ibudilast in progressive multiple sclerosis. Mult Scler. 2021 Aug;27(9):1384-1390. doi: 10.1177/1352458520964409. Epub 2020 Oct 15. PMID 33054533
- [Derived] Fox RJ, Coffey CS, Conwit R, Cudkowicz ME, Gleason T, Goodman A, Klawiter EC, Matsuda K, McGovern M, Naismith RT, Ashokkumar A, Barnes J, Ecklund D, Klingner E, Koepp M, Long JD, Natarajan S, Thornell B, Yankey J, Bermel RA, Debbins JP, Huang X, Jagodnik P, Lowe MJ, Nakamura K, Narayanan S, Sakaie KE, Thoomukuntla B, Zhou X, Krieger S, Alvarez E, Apperson M, Bashir K, Cohen BA, Coyle PK, Delgado S, Dewitt LD, Flores A, Giesser BS, Goldman MD, Jubelt B, Lava N, Lynch SG, Moses H, Ontaneda D, Perumal JS, Racke M, Repovic P, Riley CS, Severson C, Shinnar S, Suski V, Weinstock-Guttman B, Yadav V, Zabeti A; NN102/SPRINT-MS Trial Investigators. Phase 2 Trial of Ibudilast in Progressive Multiple Sclerosis. N Engl J Med. 2018 Aug 30;379(9):846-855. doi: 10.1056/NEJMoa1803583. PMID 30157388
- See also: Related Info — http://www.neuronext.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibudilast | Placebo Oral Capsule
Started | 129 | 126
Completed | 108 | 112
Not Completed | 21 | 14
Not completed — Adverse Event | 10 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Multiple sclerosis progression | 3 | 2
Not completed — Wanted to try therapy not permitted | 1 | 0
Not completed — Subject declined future visits | 0 | 1
Not completed — Left geographical area | 2 | 0
Not completed — Too many pills | 1 | 0
Not completed — MS Relapse | 0 | 1
Not completed — Chose to join a stem cell trial | 0 | 1
Not completed — Subject bedridden, rapidly declining | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibudilast | Placebo Oral Capsule | Total
Number analyzed (Participants) | 129 | 126 | 255
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 54.0 (7.8) | 56.1 (6.6) | 56.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 62 | 57 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 125 | 121 | 246
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 122 | 114 | 236
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 129 | 126 | 255

OUTCOME MEASURES:

1. Primary Outcome: Covariate-adjusted Mean Rate of Change in Brain Atrophy Over 96 Weeks as Measured by Brain Parenchymal Fraction (BPF).
Description: To evaluate the activity of ibudilast (100 mg/day) versus placebo at 96 weeks as measured by quantitative magnetic resonance imaging (MRI) analysis for whole brain atrophy using brain parenchymal fraction (BPF), calculated as the ratio of brain parenchymal tissue volume to the total volume contained within the brain surface contour.
Time Frame: 96 weeks
Population: Modified intent-to-treat is the primary population for efficacy analysis, defined as all participants from the intent-to-treat population (all participants randomly assigned) who received at least one dose of study medication, have at least one efficacy assessment for at least one primary or secondary parameter in the double-blind treatment phase.
Measure: Mean (90% Confidence Interval); unit: ratio
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 103 | 111
ratio | -0.00168 [-0.00288 to -0.00048] | -0.00392 [-0.00491 to -0.00293]
Statistical Analysis 1: Comparison: Ibudilast vs Placebo Oral Capsule; The null hypothesis states that the BPF rates of change in the treatment and placebo groups are equal, which can be evaluated based on as assessment of parameter estimates from a linear mixed model (LMM); Test type: Superiority; p = 0.04, t-test, 2 sided

2. Primary Outcome: Percentage of Participants With Adverse Events.
Description: Safety Measures: percentage of participants who experienced treatment-emergent adverse events, clinically significant abnormal laboratory and electrocardiogram results.
Time Frame: 96 weeks
Population: Safety analysis population: comprises all subjects who received at least one dose of study medication. This is the population for all safety analyses, and subjects were analyzed based on the treatment they received.
Measure: Number (90% Confidence Interval); unit: percentage receiving study medication
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 129 | 126
percentage receiving study medication | 92.2 [87.2 to 95.7] | 88.1 [82.3 to 92.5]

3. Secondary Outcome: Diffusion Tensor Imaging (DTI) in Descending Pyramidal White Matter Tracts
Description: Diffusion tensor imaging estimates the three-dimensional diffusion of water in brain tissue and has been explored as an outcome in MS.
Time Frame: 48 weeks
Population: modified intent-to-treat population
Measure: Least Squares Mean (90% Confidence Interval); unit: 10^3/mm^2/s
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 103 | 111
10^3/mm^2/s
  Left axial diffusivity mean | 0.0001 [-0.0068 to 0.0070] | -0.0006 [-0.0074 to 0.0061]
  Left radial diffusivity mean | -0.0077 [-0.0131 to -0.0023] | 0.0027 [-0.0026 to 0.0081]
  Right axial diffusivity mean | 0.0014 [-0.0055 to 0.0084] | -0.0017 [-0.0085 to 0.0051]
  Right radial diffusivity mean | -0.0029 [-0.0088 to 0.0031] | 0.0046 [-0.0012 to 0.0104]

4. Secondary Outcome: Magnetization Transfer Ratio (MTR) Imaging in Normal-appearing Brain Tissue
Description: A magnetization transfer MRI as a marker of brain myelin content including the cerebral cortex could be useful. MT imaging provides access to the restricted protons, which are located in biologically interesting tissue regions.Cortical and normal appearing grey matter MTR correlates strongly with measures of disability such as the multiple sclerosis functional composite score and can show treatment effects.
Time Frame: 96 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 95 | 103
ratio | 0.325 [0.285 to 0.365] | 0.247 [0.195 to 0.299]

5. Secondary Outcome: Retinal Nerve Fiber Layer as Measured by Optical Coherence Tomography (OCT).
Description: Mean retinal nerve fiber layer thickness from baseline measured by Optical coherence tomography (OCT), a non-invasive imaging technique used to obtain high-resolution cross-sectional images of the retina. Increase in thickness is considered improvement.
Time Frame: 96 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: micrometers
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 94 | 103
micrometers | 83.0 [80.7 to 85.2] | 79.5 [77.2 to 81.7]

6. Other Pre Specified Outcome: New T1 Lesions Since Baseline
Description: New T1 lesions since baseline as measured by least square mean (90% confidence interval).
Time Frame: 96 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: lesions
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 102 | 110
lesions | 0.355 [0.202 to 0.507] | 0.317 [0.170 to 0.463]

ADVERSE EVENTS:
Time Frame: 100 weeks
Arm/Group | Ibudilast | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/126
Serious Adverse Events (participants affected / at risk) | 20/129 | 24/126
Other Adverse Events (participants affected / at risk) | 119/129 | 111/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibudilast (N=129) | Placebo Oral Capsule (N=126)
ataxia (Nervous system disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cystitis (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
febrile neutropenia (Hepatobiliary disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 1 (1)
metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
colelithiais (Hepatobiliary disorders) | 0 (0) | 1 (1)
colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
parotidectomy (Endocrine disorders) | 0 (0) | 1 (1)
intestinal obstraction (Gastrointestinal disorders) | 0 (0) | 1 (1)
bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
kideny infection (Renal and urinary disorders) | 0 (0) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
bladder transitional cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
tooth infection (Infections and infestations) | 0 (0) | 1 (1)
convulsion (Nervous system disorders) | 0 (0) | 1 (1)
cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibudilast (N=129) | Placebo Oral Capsule (N=126)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 4 (7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 3 (3)
Conjunctivitis (Eye disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 35 (39) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 19 (21) | 8 (9)
Vomiting (Gastrointestinal disorders) | 9 (10) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (10) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (3)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Fatigue (General disorders) | 14 (14) | 10 (11)
Oedema peripheral (General disorders) | 5 (6) | 6 (6)
Irritability (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 35 (67) | 43 (88)
Upper respiratory tract infection (Infections and infestations) | 13 (17) | 24 (26)
Sinusitis (Infections and infestations) | 5 (7) | 6 (7)
Bronchitis (Infections and infestations) | 5 (5) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Tooth infection (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Influenza like illness (Infections and infestations) | 1 (1) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (10)
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 29 (63) | 20 (35)
Laceration (Injury, poisoning and procedural complications) | 6 (7) | 7 (8)
Contusion (Injury, poisoning and procedural complications) | 6 (8) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 5 (6) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Urine analysis abnormal (Investigations) | 4 (4) | 4 (4)
Hepatic enzyme increased (Investigations) | 4 (5) | 3 (4)
Lymphocyte count decreased (Investigations) | 4 (4) | 2 (2)
White blood cell count decreased (Investigations) | 4 (5) | 0 (0)
Gamma-glutamyl transferase increased (Investigations) | 4 (4) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (13) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 15 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 13 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 23 (29) | 15 (19)
Muscle spasticity (Nervous system disorders) | 9 (9) | 12 (13)
Paraesthesia (Nervous system disorders) | 9 (11) | 8 (8)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 14 (16) | 11 (11)
Depression (Psychiatric disorders) | 12 (15) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 4 (5) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 8 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Hot flush (Vascular disorders) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT01982942/Prot_SAP_ICF_000.pdf